CLINICAL TRIAL: NCT01095484
Title: Named Patient Program With Rotigotine Transdermal System
Status: Completed | Type: Observational
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: SP0953
Record Dates: First submitted 2010-03-26; First posted 2010-03-30 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2012-12

CONDITIONS: Conditions for Which There is a Documented Medical Necessity to Receive Treatment With Rotigotine
Keywords: Rotigotine; Neupro®

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Rotigotine: Patients who have a documented medical necessity to receive treatment with rotigotine treatment in accordance with standard medical practice.
  Interventions: Drug: Rotigotine patch

INTERVENTIONS:
Drug: Rotigotine patch — 1 patch daily for up to 48 months. Patch strength (per 24 hours): 1 mg - 8 mg based on investigator's assessment
  Other Names: Neupro patch

SUMMARY:
The named patient program will allow investigators to supply rotigotine transdermal system to patients who have a documented medical necessity to receive treatment with the drug.

ELIGIBILITY:
Inclusion Criteria:

* Subject is informed and given ample time and opportunity to think about her/his participation and has given her/his written informed consent
* Subject is willing and able to comply with all trial requirements
* Subject either:

  1. is currently taking no more than 3 mg/24 h Rotigotine for Idiopathic Restless Legs Syndrome (RLS) in adults, 6 mg/24 h Rotigotine for early-stage Parkinson's disease, 8 mg/24 h Rotigotine for advanced stage Parkinson's disease (ie, treated with concomitant l-dopa) and has tried and failed an adequate course of another dopamine agonist, with failure defined as either suboptimal control of symptoms or the development of intolerable Adverse Events (AEs) (eg, hallucinations), or
  2. is not taking Rotigotine but has previously demonstrated an adequate response following an appropriate course of treatment with another dopamine agonist or l-dopa, based on the investigator's assessment and has tried and failed an adequate course of another dopamine agonist, or
  3. has completed participation in UCB Rotigotine clinical trial SP0934, SP1055, or RL0003
* The investigator attests to the medical necessity of treatment with Rotigotine in contrast to alternate treatments (eg, dysphagia).
* The investigator receives written approval from the Sponsor to enroll the subject

Exclusion Criteria:

* Subject is pregnant or nursing or is of child bearing potential but (i) not surgically sterile or (ii) not using adequate birth control methods or (iii) not sexually abstinent or (iv) subject is not at least 2 years postmenopausal
* Subject has any other clinically significant medical condition, psychiatric condition, or laboratory abnormality that would, in the judgment of the investigator, interfere with the subject's ability to participate in the trial
* Subject has a lifetime history of suicide attempt (including an active attempt, interrupted attempt, or aborted attempt), or has suicidal ideation in the past 6 months as indicated by a positive response ("Yes") to either Question 4 or Question 5 of the Columbia Suicide Severity Rating Scale (C SSRS) at Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have a documented medical necessity to receive treatment with rotigotine treatment in accordance with standard medical practice.
Sampling Method: Non-Probability Sample
Enrollment: 520 (Actual)
Dates: Start 2008-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Adverse Events as reported spontaneously by the subject or as assessed by the investigator at the maintenance visits (about every three months) | From Baseline to End of Study (up to 48 months)
  Adverse events as reported spontaneously by the subject or as assessed by the investigator at the maintenance visits (about every three months)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (51):
- United States (51):
  - 088, Birmingham, Alabama
  - 082, Cullman, Alabama
  - 085, Fairhope, Alabama
  - 014, Huntsville, Alabama
  - 097, Gilbert, Arizona
  - 003, Phoenix, Arizona
  - 044, Phoenix, Arizona
  - 036, Berkeley, California
  - 024, Fountain Valley, California
  - 034, Irvine, California
  - 019, Los Angeles, California
  - 040, Orange, California
  - 076, Sunnyvale, California
  - 035, Fort Collins, Colorado
  - 027, Washington D.C., District of Columbia
  - 070, Atlantis, Florida
  - 002, Boca Raton, Florida
  - 031, Clearwater, Florida
  - 028, Largo, Florida
  - 075, Ormond Beach, Florida
  - 022, St. Petersburg, Florida
  - 004, Tampa, Florida
  - 054, Weston, Florida
  - 030, Atlanta, Georgia
  - 041, Honolulu, Hawaii
  - 011, Peoria, Illinois
  - 025, Destrehan, Louisiana
  - 091, Clinton Township, Michigan
  - 001, Southfield, Michigan
  - 042, Warren, Michigan
  - 037, Ocean Springs, Mississippi
  - 016, West Plains, Missouri
  - 026, Lincoln, Nebraska
  - 086, Freehold, New Jersey
  - 062, Ridgewood, New Jersey
  - 018, Albany, New York
  - 066, Brooklyn, New York
  - 006, Patchogue, New York
  - 052, Charlotte, North Carolina
  - 093, Salisbury, North Carolina
  - 065, Albany, Oregon
  - 009, Salem, Oregon
  - 048, Austin, Texas
  - 072, Austin, Texas
  - 071, Dallas, Texas
  - 046, Houston, Texas
  - 005, Kirkland, Washington
  - 017, Olympia, Washington
  - 012, Spokane, Washington
  - 053, Tacoma, Washington
  - 056, Milwaukee, Wisconsin